CLINICAL TRIAL: NCT05219188
Title: PErirenal Adipose Tissue and RenaL Hemodynamics in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: PEARL-HFPEF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, A.A.Voors, Principal Investigator, University Medical Center Groningen
Other Study IDs: NL78282.042.21
Record Dates: First submitted 2021-12-15; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Obesity; Renal Insufficiency
MeSH Terms: conditions — Obesity; Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — spot urinary samples and 24-hours collection urinary samples EDTA-plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Heart failure with preserved ejection fraction and BMI <25: Subjects will undergo DCE-CT. Radiation exposure has been calculated to be 3.7 mS, Iomeron dose admission during CT is 50 mL containing 714 mg/ml iomeprol
  Interventions: Radiation: 3.7 mS, CT radiation
- Heart failure with preserved ejection fraction and BMI >30: Subjects will undergo DCE-CT. Radiation exposure has been calculated to be 3.7 mS, Iomeron dose admission during CT is 50 mL containing 714 mg/ml iomeprol
  Interventions: Radiation: 3.7 mS, CT radiation
- Healthy controls with BMI <25: Subjects will undergo DCE-CT. Radiation exposure has been calculated to be 3.7 mS, Iomeron dose admission during CT is 50 mL containing 714 mg/ml iomeprol
  Interventions: Radiation: 3.7 mS, CT radiation
- Healthy controls with BMI >30: Subjects will undergo DCE-CT. Radiation exposure has been calculated to be 3.7 mS, Iomeron dose admission during CT is 50 mL containing 714 mg/ml iomeprol
  Interventions: Radiation: 3.7 mS, CT radiation

INTERVENTIONS:
Radiation: 3.7 mS, CT radiation — Subjects will undergo dynamic contrast enhanced CT with an estimated radiation exposure of 3.7 mS

SUMMARY:
Rationale: Perirenal adipose tissue (PRAT) thickness has been associated to worsening renal function and hypertension. The role of PRAT in heart failure with a preserved ejection fraction (HFpEF) has never been established. The hypothesis of this study is that in patients with HFpEF the diameter of PRAT is increased compared with age, sex and BMI matched controls.

Objective: The main objective is to determine whether PRAT thickness is increased in patients with HFpEF. Secondary objectives are to determine whether PRAT thickness is correlated to whole kidney perfusion, renal venous flow patterns, markers of glomerular and tubular damage and dysfunction, NT pro-BNP, renin and aldosterone. Lastly, this study aims to determine whether these correlations are similar for men and women with HFpEF.

Study design: the proposed study is a single center, cross-sectional observational case-control study, including 30 HFpEF patients and 30 healthy controls.

Study population: Adult patients with HFpEF with a body mass index (BMI) of <25.0 or >30.0 and healthy age, sex and BMI-matched controls.

Intervention (if applicable): Not applicable. Main study parameters/endpoints: The primary endpoint will be the difference in diameter and volume of perirenal adipose tissue measured on dynamic contrast computed CT (DCE-CT) in patients with HFpEF vs. healthy age, sex and BMI matched controls.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participating subjects will be asked to visit the University Medical Center Groningen (UMCG) twice (once for screening, once for testing visit). During the testing visit they will undergo intravenous contrast abdominal CT, renal sonography, blood drawing and urine collection. Risks associated with these procedure are very limited, rare and include bleeding and infection for venapunction, and contact dermatitis for ultrasound gel. Adverse events for CT include hypersensitivity reactions to contrast agent, which include skin rash, hypotension and bronchospasm.

ELIGIBILITY:
Inclusion criteria (patient category):

1. Able and willing to give written informed consent
2. Male and female subjects with age >18 years
3. A diagnosis of HFpEF based on typical symptoms (and/or signs), a LVEF >50% (assessed within 12 months prior to baseline testing) and at least two of the following criteria10:

   1. For BMI <35.0 kg/m2: NT pro-BNP ≥220 pg/mL For BMI ≥35.0 kg/m2: NT pro-BNP ≥125 pg/mL
   2. Left atrial volume index >34 ml/m2 or Left ventricular mass index >115g/m2 (men) or >95g/m2 (women)
   3. E/e' ≥13 or e' average <9 cm/s
4. BMI <25 or >30

Exclusion criteria for patient category:

1. Amyloid cardiomyopathy or cardiomyopathy due to sarcoïdosis or M. Fabry, as reflected by medical history.
2. Atrial fibrillation on ECG performed at screening
3. Genetic hypertrophic (obstructive) cardiomyopathy.
4. Severe (grade III/III) aortic stenosis.
5. Female patient with childbearing potential, aiming to get pregnant or pregnant at the time of inclusion.
6. Patients on (intermittent or continuous) hemodialysis
7. Proven hypersensitivity to iodine contrast or any other contra-indication for computed tomography.

Inclusion criteria for healthy controls:

1. Able and willing to give written informed consent
2. Male and female subjects with age >18 years
3. BMI <25 or >30

Exclusion criteria for healthy controls:

1. Diagnosis of any cardiovascular disease, either in the medical history or diagnosed during screening.
2. Diagnosis of diabetes mellitus, defined as use of glucose lowering drugs
3. Diagnosis of hypertension, defined as mean of 3 blood pressures measurements of >140/90 mmHg at screening or use of blood pressure lowering drugs.
4. Female patients with childbearing potential, either already pregnant or aiming to get pregnant at the time of inclusion.
5. Proven hypersensitivity to iodine contrast or any other contra-indication for computed tomography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic, stable HFpEF with and without obesity will be compared to healthy controls with and without obesity.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Perirenal fat thickness | Up to 28 days after screening
  The primary objective is to determine whether perirenal adipose tissue thickness is increased in patients with HFpEF compared with age, sex and BMI-matched healthy controls

SECONDARY OUTCOMES:
Kidney perfusion | Up to 28 days after screening
  Determine whether a greater PRAT volume correlates to impaired kidney perfusion on DCE- CT in patients with HFpEF
Renal venous flow patterns | Up to 28 days after screening
  Determine whether a greater PRAT volume correlates to renal venous flow patterns assessed with ultrasound in patients with HFpEF
eGFR on CDE-CT | Up to 28 days after screening
  Determine whether a greater PRAT volume correlates to glomerular filtration rate assessed with CDE- CT.
Renal biomarkers | Up to 28 days after screening
  Determine whether a greater PRAT volume correlates to markers of glomerular and tubular damage and dysfunction (urinary KIM-1, urinary OPN, serum creatinine, plasma Cystatin C) in patients with HFpEF
Heart failure severity | Up to 28 days after screening
  Determine whether a greater PRAT volume correlates to plasma NT pro-BNP, renin and aldosterone concentrations in patients with HFpEF as well as to pulmonary arterial pressure as assessed with cardiac ultrasound.
Sex differences | Up to 28 days after screening
  Determine whether correlations between renal hemodynamics and PRAT volumes are different between men and women with HFpEF.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan A Voors, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang N, Mao EW, Hou NN, Liu YP, Han F, Sun XD. Novel insight into perirenal adipose tissue: A neglected adipose depot linking cardiovascular and chronic kidney disease. World J Diabetes. 2020 Apr 15;11(4):115-125. doi: 10.4239/wjd.v11.i4.115. PMID 32313610
- [Result] Jeong S, Park SB, Chang IH, Shin J, Chi BH, Park HJ, Lee ES. Estimation of renal function using kidney dynamic contrast material-enhanced CT perfusion: accuracy and feasibility. Abdom Radiol (NY). 2021 May;46(5):2045-2051. doi: 10.1007/s00261-020-02826-7. Epub 2020 Oct 22. PMID 33090257
- [Result] Sun X, Han F, Miao W, Hou N, Cao Z, Zhang G. Sonographic evaluation of para- and perirenal fat thickness is an independent predictor of early kidney damage in obese patients. Int Urol Nephrol. 2013 Dec;45(6):1589-95. doi: 10.1007/s11255-013-0404-4. Epub 2013 Mar 6. PMID 23463155